CLINICAL TRIAL: NCT03957863
Title: Study of Erythropoietin in Newborns and Children
Acronym: EPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Girodon 2018
Record Dates: First submitted 2019-05-15; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Newborn Infant; Child Under One Year of Age
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Plasma collection for EPO assay — Plasma collection for EPO assay

SUMMARY:
Erythropoietin (EPO) is a glycoprotein hormone with a molecular weight of 30.4 kDa, responsible for regulating erythropoiesis in adults, newborns and fetuses. During pregnancy, the concentration of maternal serum EPO increases linearly to allow for effective erythropoiesis over time. In the fetus, in the first 30 weeks of gestation, the liver is the main synthetic organ. Thereafter, there is a progressive transfer of the synthesis of EPO to the kidneys. In the long term, under normal conditions of oxygenation, the fetal synthesis of EPO is mainly ensured by the kidney.

Because of the impossibility of making EPO tissue reserves and the inability of EPO to pass the placental barrier, the concentration of circulating EPO in the fetus reflects the balance between production and elimination. During the last trimester of pregnancy, in the absence of patent hypoxia, fetal concentrations of circulating EPO are between 10 and 50 mIU /ml, while in amniotic fluid the EPO is found at lower concentrations, between 2 and 20 mIU /ml.

In adults, EPO synthesis is primarily renal, and incidentally hepatic, even if in certain pathological situations (end-stage kidney disease or polycystosis) the liver is able to take over and synthesize EPO with an electrophoretic profile similar to that of the EPO from the umbilical cord, but often in insufficient quantities.

The objective of this study is to describe the forms of EPO in newborns and to compare possible iso-forms with those of adults.

ELIGIBILITY:
Inclusion Criteria:

* infant or child under 1 year old hospitalized or consulting at CHU Dijon Bourgogne whose parents have not opposed participation in the study

Exclusion Criteria:

* child treated with recombinant erythropoietin

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborn or child under 1 year of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
EPO concentration UI/L | Baseline
Electrophoretic profile of EPO | Baseline
  It is an indicator of glycosylation differences (more complex forms including sialic acids are more acidic, less complex forms are more basic)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Derived] Martin L, Maric D, Idriss S, Delamare M, Le Roy A, Maaziz N, Caillaud A, Si-Tayeb K, Robriquet F, Lenglet M, Erceau L, Bellanne-Chantelot C, Plo I, Aral B, Garrec C, Airaud F, Gianfermi C, Antunes V, Keppner A, Vincent SM, Desfontaine A, Mode N, Laporte F, Gaignerie A, Chariau C, Leray I, Rogue C, David L, Redon R, Bezieau S, Mansour-Hendili L, Galacteros F, Maillet T, Pasquet M, Cougoul P, Nloga AM, Gardin C, Guitton C, Dubruille V, Giacobbi-Milet V, Leblanc T, Kaya Z, Semama D, James C, Carillo S, Ochmann M, Waage A, Mortier E, Maillasson M, Quemener A, Cario H, Skoda RC, Zermati Y, Hoogewijs D, Marchand A, Girodon F, Gardie B. Identification of Hepatic-like EPO as a Cause of Polycythemia. N Engl J Med. 2025 May 1;392(17):1684-1697. doi: 10.1056/NEJMoa2414954. PMID 40305710